CLINICAL TRIAL: NCT02855593
Title: Exploring Patient and Physician Experiences of Medical Acupuncture
Acronym: APPE
Status: Active, not recruiting | Type: Observational
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FWH20160066H
Record Dates: First submitted 2016-07-27; First posted 2016-08-04 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Attitudes
Keywords: acupuncture
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Physicians: Physicians who perform acupuncture
- Patients: Patients who have received acupuncture treatment in the past

SUMMARY:
The proposed qualitative inquiry seeks to understand medical acupuncture from both the physician and the patient perspective. Interviewees will be asked to describe their experiences from the point of diagnosis or training up until the present day to capture the nature of their experiences across the treatment trajectory. Sample size for the qualitative data collection will be based on saturation of themes (thematic findings, e.g., patient talk is limited by family knowledge or physician-patient communication is limited by time constraints in the clinical setting), meaning investigators will continue recruitment until they are no longer hearing new experiences from participants. Saturation will be kept separate by groups (i.e., saturation of themes must be met within the group of patients separately from providers). Investigators will conduct preliminary data analysis after each 10 interviews to determine when saturation is reached. Recruitment numbers here are anticipated maximum numbers needed to reach saturation. Investigators plan to recruit and sample provider and patient populations in the following way. Investigators will group physicians by the physician's training so that we are sensitive to the fact that helpful patient-physician interaction approaches may differ across the patient's lifespan or with patient or physician experience with acupuncture. Audio recordings from each interview will be professionally transcribed and analysis will be concurrent with data collection to ensure reliability and validity of findings. Investigators will review transcripts as data are collected to identify emergent themes and ensure thematic saturation.

DETAILED DESCRIPTION:
Investigators will obtain signed Informed Consent Document and HIPAA Authorization. During the screening process, data will be gathered about race, ethnicity, gender, history, and satisfaction rating of prior acupuncture received, and whether or not acupuncture has decrease reliance on prescription and over-the-counter medication use via the Screening Tool. Acknowledging the clinical partnership of patient and provider, the proposed qualitative inquiry seeks to understand medical acupuncture from both the physician and the patient perspective. A modified version of two interview techniques [Lifeline Interview Method (LIM) and Retrospective Interview Technique (RIT)] will be used. From this approach, narrative data can be analyzed both quantitatively and qualitatively and provide a visual depiction across time. In the RIT method, each participant receives a modified version of an RIT graph before the interview. The graph provides participants time to reflect on their experiences and behavior. The interviews will all be one-on-one interviews and will take approximately 90 minutes for each group, including the time for completing the RIT graph during the interview.

Interviewees will be asked to describe their experiences from the point of diagnosis or training up until the present day to capture the nature of their experiences across the treatment trajectory. Questions will address the nature of their experiences beginning with the first time the provider introduced acupuncture to the patient and up to the present day to elicit rich details about the impact of acupuncture on their social/relational lives as well as perceived psychological and physical health. Questions will also be centered on the role of communication in facilitating receptivity and adherence to an acupuncture treatment plan both in terms of provider-patient interaction and patients' interactive experiences within their social network. For physicians, questions will address pre-training and post-training perceptions of acupuncture as well.

Ultimately, the impact of acupuncture on patients' lives will be examined using the "turning point" approach. By centering on turning points individuals have the opportunity to reflect on notable moments of change that are memorable because of their impact on health, health behavior as well as health perceptions. Such turning points can also be helpful in identifying challenges patients and their physicians face with regard to adopting and adhering to acupuncture treatment. In this approach participants consider how the treatment impacted their life across time as they plot changes ("turning points") that emerged across the treatment trajectory. Time will be represented on the horizontal axis of the graph, while impact of acupuncture (as is perceived by the participant) will be represented on the vertical axis. Impact of treatment will be considered as changes that capture how treatment has a positive effect (enhancing health, enhancing receptivity, or adherence) or negative (inhibiting health, not facilitating receptivity or adherence). These turning points are always communicatively managed and, thus, the communicative nature will give rise to communication factors that facilitate the treatment and health-promoting outcomes as well as barriers (and thus, contribute to the treatment not being perceived as beneficial). From this approach, participants use a visual tool (turning point graph) to plot turning points. Once completed they connect the points with a line to provide a trajectory that illustrates how the treatment impacted their lives across the acupuncture treatment (patients) or how the treatment impacted the lives of their patients (providers).

This interview technique helps facilitate a storied approach for the participants sharing their insider experiences thereby facilitating disclosure in a more natural manner and generating narrative data rich for intervention-making. This approach allows for a translational approach to research as the narratives can be used to develop interventions and medical education critical for facilitating this form of care.

Sample size for the qualitative data collection will be based on saturation of themes (thematic findings, e.g., patient talk is limited by family knowledge or physician-patient communication is limited by time constraints in the clinical setting, meaning investigators will continue recruitment until investigators are no longer hearing new experiences from participants. Saturation will be kept separate by groups (i.e., saturation of themes must be met within the group of patients separately from providers). Generally saturation is met with 10-30 individuals within a group, depending upon how diverse the groups are (other demographic variables may require more participants and an amendment to increase the approved number of enrollments). Investigators plan to recruit and sample provider and patient populations in the following way.

Since investigators are concerned with communication differences based on training maturity, investigators will group physicians by the physician's training so that investigators are sensitive to the fact that helpful patient-physician interaction approaches may differ across the lifespan or with experience. Our goal is to interview physicians who are just completing training and physicians who completed training more than three years prior. Thus, investigators will have a "newly trained" provider group and an "experienced" provider group. For each group, investigators will ask them about the entirety of their experiences (from the point of training up to the present day) and analyze that data about patient-physician communication according to the training phase of the physician. This will ensure investigators have both in-the-moment reflections about experiences and retrospective accounts. For patients, investigators will recruit 2 groups: those seeking treatment for either 1) chronic or 2) acute conditions. Given gendered differences in health behavior and perceptions, investigators will aim to have representative male and female populations within each group.

Audio recordings from each interview will be professionally transcribed and analysis will be concurrent with data collection to ensure reliability and validity of findings. Professional transcriptionists will complete transcription of pseudoanonymous recordings. Investigators will review transcripts as data are collected to identify emergent themes and ensure thematic saturation. Qualitative data will be analyzed according to van Manen's"selective approach," using the software program ATLAS.ti.to manage large data sets. Three analytical steps according to the constant comparative method and outlined by Strauss and Corbin will be employed, beginning with the discovery of concepts and assignment of codes to text. The thematic analysis then proceeds with identifying categories by grouping related concepts to reach "thematic salience," as reflected in recurrence, repetition, and forcefulness. The final step involves defining themes and dimensions of these categories to ensure thick description. Separate analyses will be conducted for each research question and for each group and then compared across groups. Investigators will incorporate final sets of themes into action-oriented thematic statements using Banning's ecological sentence synthesis approach to ensure the research can be more easily translated into practice. These action-oriented statements can more easily be integrated into interventions and psychosocial materials in an effort to enhance provider-patient communication and shared decision making, the health care system, and by offering patients and physicians a roadmap of barriers that might impede care practice or patient adherence as well as communication strategies that can facilitate and enhance acupuncture treatment (both for patients and providers).

ELIGIBILITY:
Inclusion:

* Male and female Department of Defense beneficiaries, age 18 years or older, who have received acupuncture OR
* Male and female acupuncture providers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female Department of Defense beneficiaries ages 18 years or older who have received acupuncture and Male and female acupuncture providers will be recruited at the Mike O'Callaghan Federal Medical Center (MOFMC). No special populations (e.g., pregnant women, children, prisoners, detainees) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Retrospective Interview Technique | one year

SECONDARY OUTCOMES:
Lifeline Interview Method | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Clark, MBA/HCM, Principal Investigator — Mike O'Callaghan Federal Medical Center
Locations (1):
- Mike O'Callaghan Federal Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
no plans to share data